CLINICAL TRIAL: NCT04422379
Title: COVID-19 and Liver Injury in Patients With or Without Underlying Liver Disease: A Multi-centre Retrospective-prospective Observational Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Max Healthcare Insititute Limited (Other)
Responsible Party: Sponsor
Other Study IDs: COVID 19/LI/2020
Record Dates: First submitted 2020-06-07; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID-19 and liver injury in patients with or without underlying liver disease: A multi-centre retrospective-prospective observational study.

All patients infected with SARS-CoV-2 and admitted to the COVID-19 ward/ICU of Max Hospital Saket (either in East Wing , Max Super Specialty Hospital, Saket or MAX Smart Super Specialty Hospital, Saket) between 1/4/2020 to 30/6/2020 (retrospective data between 1/4/2020- 30/5/2020 & prospective data from approval till 30/6/2020), will be included

DETAILED DESCRIPTION:
COVID-19 and liver injury in patients with or without underlying liver disease: A multi-centre retrospective-prospective observational study.

All patients infected with SARS-CoV-2 and admitted to the COVID-19 ward/ICU of Max Hospital Saket (either in East Wing , Max Super Specialty Hospital, Saket or MAX Smart Super Specialty Hospital, Saket) between 1/4/2020 to 30/6/2020 (retrospective data between 1/4/2020- 30/5/2020 & prospective data from approval till 30/6/2020), will be included Primary objectives

1. To study the prevalence of liver live injury & factors associated with among patients in-fected with SARS-CoV-2.
2. To study the prevalence of new liver injury and factors associated with it, among patient with underlying liver disease who develops COVD-19.

Secondary objectives

1. To correlate the presence and degree of liver dysfunction with the clinical outcomes in these patients.
2. To define the incidence of development of acute liver failure among these patients

ELIGIBILITY:
Inclusion Criteria:All patients infected with SARS-CoV-2 and admitted to the COVID-19 ward/ICU of Max Hospital Saket (either in East Wing , Max Super Specialty Hospital, Saket or MAX Smart Super Specialty Hospital, Saket) between 1/4/2020 to 30/6/2020 (retrospective data between 1/4/2020- 30/5/2020 & prospective data from approval till 30/6/2020), will be included.

-

Exclusion Criteria:

1. Patients less that 18 years old with COVID-19
2. Pregnant ladies with COVD-19
3. Unwilling to give consent for inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include all the COVID 19 patients (male & female) with minimum age 18 years old. And take 60% patient in Retrospective arm and 40% patient in prospective arm.
Sampling Method: Probability Sample
Enrollment: 314 (Estimated)
Dates: Start 2020-06-07 (Estimated); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
COVID-19 Positive Case | 4-8 weeks
  To study the prevalence of liver live injury & factors associated with among patients in-fected with SARS-CoV-2.
COVID-19 Positive Case | 4-8 weeks
  To study the prevalence of new liver injury and factors associated with it, among patient with underlying liver disease who develops COVID-19.

SECONDARY OUTCOMES:
COVID-19 Positive Case | 4-8 weeks
  To correlate the presence and degree of liver dysfunction with the clinical outcomes in these patients.
COVID-19 Positive Case | 4-8 weeks
  To define the incidence of development of acute liver failure among these patients

CONTACTS AND LOCATIONS:
Overall Officials: Kaushal Madan, DM, Principal Investigator — Max healthcare
Locations (1):
- Max Super Speciality Hospital, Saket (A Unit Of Devki Devi Foundation), New Delhi, Dlelhi, India

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing protocol is undecided at this stage. We may, however, provide the data if requested.